CLINICAL TRIAL: NCT01420835
Title: Randomized Clinical Trial: Chinese Auriculotherapy With and Without Protocol on Stress and Quality of Life in Nursing Professionals
Brief Title: Chinese Auriculotherapy on Stress and Quality of Life in Nursing Professionals: Randomized Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Sociedade Hospital Samaritano (Other)
Responsible Party: Principal Investigator, Leonice Fumiko Sato Kurebayashi, Leonice Fumiko Sato Kurebayashi, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SISNEP CAAE 0050.0.196.196-11
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Stress; Quality of Life
Keywords: Stress; Quality of life
MeSH Terms: interventions — Auriculotherapy; Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Without Protocol Group (Active Comparator): The chinese auriculotherapy is a intervention used by Chinese Traditional Medicine in order to balance the body energy and to treat several kind of diseases using semi-permanent needles in specific points of the auricular pavilion.
  Five points will be chosen to treat stress according to the symptoms and Chinese diagnosis.
  Interventions: Other: without protocol group
- Auriculotherapy with protocol (Active Comparator): Auriculotherapy with stress protocol points. Five points are indicated for stress (Liver yang1, Liver yang2, Shenmen, Brainstem and Kidney).
  Interventions: Other: Auriculotherapy (protocol group)
- Control Group (No Intervention): Control Group won't receive any treatment and will be evaluated at the same time and the same way of interventions group

INTERVENTIONS:
Other: Auriculotherapy (protocol group) — The auriculotherapy points of the protocol group will be 5 points (Liver yang1, Liver yang2, Shenmen, Kidney, Brainstem), during 45 days, twice per week, 12 sessions and assessment of the follow-up (30 days) after finishing the treatment.
  Other Names: auricular acupuncture
  Arms: Auriculotherapy with protocol
Other: without protocol group — The chinese auriculotherapy is a intervention used by Chinese Traditional Medicine in order to balance the body energy and to treat several kind of diseases using semi-permanent needles in specific points of the auricular pavilion. Five points will be chosen to treat stress according to the symptoms and the Chinese diagnosis.
  Other Names: auricular acupuncture
  Arms: Without Protocol Group

SUMMARY:
The purpose of this study is to assess stress levels and quality of life in the nursing team of Samaritan Hospital and evaluate the effectiveness of Chinese auriculotherapy used with and without closed protocol on reducing the stress levels and improvement of life quality.

DETAILED DESCRIPTION:
Based on the positive results achieved in a preliminary study conducted in January and February 2010, entitled "Applicability of auricular needles or seeds for the reduction of stress in nursing professionals" at the University Hospital, emerged from this research project in order to extend the first study, with a more representative sample and with a design that would allow further discussions on the effectiveness of Chinese auricular needles semi-permanent to reduce stress and thereby improving the quality of life of nursing professionals. This clinical trial aims, above all, compare the results of the technique with the use of closed protocol and a group without protocol. The latter, however, shall be based on energy evaluation according to Traditional Chinese Medicine (TCM) and the course of treatment will be performed similarly to the clinical practice commonly performed by traditional practitioners, that is, individually, not necessarily repetitive and whose continuation is achieved depending on the answers to each treatment.

Discussions are justified about protocol and no protocol research in complementary and integrative practices, since the methodologies proposed and accepted by the scientific community does not always seem to be appropriate tools for evaluating therapies like those coming from the East. The transfer of the Western conception of research according to positivist principles are not always consistent with the principles underlying the complementary and alternative therapies, and in particular the practice from China.

ELIGIBILITY:
Inclusion Criteria:

Score by the List of Stress Symptoms (40 to 95 points)

Voluntary participation in the study

Availability of time for submission to the sessions

Exclusion Criteria:

Pregnancy

Medical license or vacation during the period

If they perform another chinese treatment like a massage, acupuncture, moxibustion etc

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
stress levels | 75 days
  The measurement of stress levels will be performed by List of Stress Symptoms (Vasconcellos) and the main symptoms

SECONDARY OUTCOMES:
quality of life domains | 75 days
  The assessment of life quality domains will be done by SF36v2

CONTACTS AND LOCATIONS:
Overall Officials: Leonice FS Kurebayashi, Principal Investigator — Instituto de Terapia Integrada e Oriental
Locations (1):
- Samaritan Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Giaponesi ANL, Leão ER. Auriculotherapy as an intervention to reduce stress reduction among the nursing team in intensive care. Nursing (São Paulo);12(139):575-579, dez. 2009. ilus.
- [Derived] Kurebayashi LF, Silva MJ. Efficacy of Chinese auriculotherapy for stress in nursing staff: a randomized clinical trial. Rev Lat Am Enfermagem. 2014 May-Jun;22(3):371-8. doi: 10.1590/0104-1169.3239.2426. PMID 25029046